CLINICAL TRIAL: NCT06388109
Title: Randomized Control Trial of Positive Peers mHealth App as a Clinic-based Intervention to Optimize HIV Outcomes Among Young, Minority Persons Living With HIV
Brief Title: Positive Peers Intervention Clinical Trial
Acronym: PoPIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Kent State University (Other)
Responsible Party: Principal Investigator, Ann Avery, co-Principal Investigator, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB15-00741
Record Dates: First submitted 2024-04-22; First posted 2024-04-29 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: randomized control trial with observational cohort for eligible patients who decline participation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Immediate Start (Experimental): Participants in the immediate start arm will download and begin use of the Positive Peers app at the enrollment visit.
  Interventions: Other: Positive Peers mobile app
- Delayed Start (Active Comparator): Participants in the delayed start arm will download and begin use of the Positive Peers app 6 months after enrollment
  Interventions: Other: Positive Peers mobile app
- Observational Cohort (No Intervention): Participants in the observational cohort have declined participation in the clinical trial but agree to do the baseline survey and have medical outcomes data recorded.

INTERVENTIONS:
Other: Positive Peers mobile app — Positive Peers is a multifunctional mobile app using a mind, body, spirit theme aimed to improve HIV care outcomes.
  Arms: Delayed Start; Immediate Start

SUMMARY:
The goal of this clinical trial is to learn if the Positive Peers mobile app intervention increases rates of viral suppression in young (13-34 y/o) persons with HIV.

Does use of the Positive Peers app improve viral suppression among young minority persons with HIV? What user characteristics are associated with a) viral suppression, b) retention in care, and c) perceived HIV-related stigma?

Participants will:

* download the mobile app onto their personal smartphone
* Use the mobile app as they find useful
* complete online surveys at enrollment, 3 mo, 6, mo, 9 mo and 12 months.

DETAILED DESCRIPTION:
Participants will load the Positive Peers app on their personal device (either immediately or after a 6 month delay) and be encouraged to use the app regularly. Eligible patients who decline participation in the intervention will be asked to participate in an observational arm.

All participants will complete a brief baseline survey. Participants in the immediate or delayed arms will also complete surveys at 3, 6, 9, and 12 months. Medical data will be collected from the medical record and usage data will be collected from the app itself. Medical data will be collected for 12 months prior to enrollment and 18 months after enrollment. At the end of the study, participants are welcome to continue to use the app.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* Identifies as either a racial, ethnic, sexual or gender minority

One of the following:

* Newly diagnosed within last 12 months
* Out of care (greater than 6 months between any two HIV provider visits in last 24 months)
* Not virally suppressed (any viral load > 200 copies in last 24 months)
* Has a working smartphone
* Functional English ability

Exclusion Criteria:

* prior use of Positive Peers mobile app

Ages: 13 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Viral suppression | 6 months
  Proportion of participants who have HIV viral load <200 copies/ ml

SECONDARY OUTCOMES:
Correlates of app use and viral suppression | 6 months
  Identify participant demographic and psychosocial factors from the baseline survey that correlate with app use and viral suppression (viral load < 200 copies/ ml).
Correlates of app use and retention in care | 12 months
  Identify participant demographic and psychosocial factors from the baseline survey that correlate with app use on retention in care (completing office visit at least every 6 months)
Correlates of app use and HIV related perceived stigma | 3 months
  Identify participant demographic and psychosocial factors from the baseline survey that correlate with app use and changes in HIV-related perceived stigma on the HIV Stigma scale (Eriksson).

CONTACTS AND LOCATIONS:
Overall Officials: Ann Avery, MD, Principal Investigator — MetroHealth/ CWRU; Mary Step, PhD, Principal Investigator — Kent State University
Locations (6):
- United States (6):
  - Northeast Valley Health Corporation, Van Nuys, California
  - Infectious Disease Practice- Rutgers University, Newark, New Jersey
  - Equitas Health, Cincinnati, Ohio
  - Equitas Health, Columbus, Ohio
  - Thomas Street Clinic, Houston, Texas
  - UW Madison Clinic at Harborview, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Participant survey data, backend usage data and medical record data will be deidentified and made available to researchers with a reasonable request and plan for use.
Supporting Information: Study Protocol
Time Frame: within 1 year after award ends
Access Criteria: Request for data to reproduce results or for meta-analysis.

REFERENCES:
- [Background] Step MM, McMillen Smith J, Lewis SA, Avery AK. Using the Positive Peers Mobile App to Improve Clinical Outcomes for Young People With HIV: Prospective Observational Cohort Comparison. JMIR Mhealth Uhealth. 2022 Sep 28;10(9):e37868. doi: 10.2196/37868. PMID 36170001
- [Background] Comulada WS, Step M, Fletcher JB, Tanner AE, Dowshen NL, Arayasirikul S, Keglovitz Baker K, Zuniga J, Swendeman D, Medich M, Kao UH, Northrup A, Nieto O, Brooks RA; Special Projects Of National Significance Social Media Initiative Study Group. Predictors of Internet Health Information-Seeking Behaviors Among Young Adults Living With HIV Across the United States: Longitudinal Observational Study. J Med Internet Res. 2020 Nov 2;22(11):e18309. doi: 10.2196/18309. PMID 33136057
- [Background] Step MM, Knight K, McMillen Smith J, Lewis SA, Russell TJ, Avery AK. Positive Peers Mobile Application Reduces Stigma Perception Among Young People Living With HIV. Health Promot Pract. 2020 Sep;21(5):744-754. doi: 10.1177/1524839920936244. Epub 2020 Aug 6. PMID 32757838
- [Background] Step MM, McMillen Smith J, Kratz J, Briggs J, Avery A. "Positive Peers": Function and Content Development of a Mobile App for Engaging and Retaining Young Adults in HIV Care. JMIR Form Res. 2020 Jan 30;4(1):e13495. doi: 10.2196/13495. PMID 32012035